## **INFORMED CONSENT FORM**

| I have been invited to participate in research | arch about ": Effect of repetitive binemispheric anodal transcranial |
|---|---|
| Direct Current Stimulation on motor fun | ction of patients with Parkinson's Disease". I have read the foregoing |
| information, or it has been read to me. I | have had the opportunity to ask questions about it and any questions I |
| have asked have been answered to my sa | tisfaction. I consent voluntarily to be a participant in this study. |
| Name of Participant: | |
| Signature of Participant: | |
| Date: | |
| | Day/month/year |
| If illiterate: | |
| I have witnessed the accurate reading of | the consent form to the potential participant, and the individual has had |
| the opportunity to ask questions. I confir | m that the individual has given consent freely. |
| Name of witness: | Thumb print of participant |
| Signature of witness: | |
| Date: | |
| Day | y/month/year |

## Statement by the researcher/person taking consent

I have accurately read out the information sheet to the potential participant, and to the best of my ability made sure that the participant understands that the following will be done:

1. Detailed history and physical examination will be done.

| $\sim$ | TD | 1 1 | | | | *11 | 1 1 |
|--------|-------------|----------|---------|-------|--------|------|---------|
| 2 | Transcrania | l direct | current | stimu | lation | WILL | be done |

I confirm that the participant was given an opportunity to ask questions about the study, and all the questions asked by the participant have been answered correctly and to the best of my ability. I confirm that the individual has not been coerced into giving consent, and the consent has been given freely and voluntarily. Individual has every right to opt out of this study at any point.

| Name of Researcher/person taking the consent |
|----------------------------------------------------|
| Signature of Researcher /person taking the consent |
| Date |

A copy of this ICF has been provided to the participant.